CLINICAL TRIAL: NCT06692881
Title: Evaluation of Function And Satisfaction of UbrogepanT-treated Migraine Patients in Canada (FAST): Prospective, Observational, Real-world Study
Brief Title: Study to Assess Function and Satisfaction of Oral Ubrogepant in Adult Participants After Multiple Migraine Attacks In Canada
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-245
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Migraine; ubrogepant; Ubrelvy
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ubrogepant: Participants will receive Ubrogepant as prescribed by their physician in routine clinical practice.

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will evaluate function and satisfaction with oral ubrogepant in treating adult participants after multiple migraine attacks.

Ubrogepant is a drug approved for the acute treatment of migraine in adults. Approximately 167 participants will be enrolled in approximately 10-15 sites across Canada.

Participants will receive ubrogepant as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 12 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants able to give voluntary informed consent before starting any study-related assessments or procedures (to be obtained/documented as per local regulations).
* Adults (≥18 years of age) at time of informed consent.
* Participants with at least 1-year history of migraine with or without aura consistent with a diagnosis according to the ICHD-3 (2018).
* Participants with history of experiencing at least 3 migraine attacks per month with moderate to severe symptoms
* Participants prescribed ubrogepant by investigator for the acute treatment of migraine according to local product label, independent of and prior to study participation
* Participants willing and able to comply with the requirements of the study.
* Participants with access to an electronic device (mobile phone, tablet, laptop, etc.) with internet access.

Exclusion Criteria:

* Participants previously exposed to a ubrogepant or rimegepant as routine therapy or through a clinical trial.
* Participants with history of known contraindications to ubrogepant as per local labeling.
* Participants Pregnant or planning to be pregnant or of childbearing potential not using contraception
* Participants enrolled in any interventional studies that may include investigational compounds for migraine or non-AbbVie observational studies.
* History or current evidence of any condition that might interfere with their ability to comply with the study requirements, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants receiving ubrogepant per routine clinical care for the treatment of migraine in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Functional Disability Scale (FDS) Score of =0, no disability, able to function normally 4 hours post-dose | Up to approximately 12 weeks
  Functional Disability Scale (FDS) is a Patient-Reported Outcome (PRO) assessing the ability of a participant to perform daily activities, rated on a 4-point scale (0=no disability, able to function normally; to 3=severely impaired, cannot do all or most things, bed rest may be necessary)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Canada (13):
  - Calgary Headache Assessment and Management Program /ID# 271475, Calgary, Alberta
  - Burrard Health Center /ID# 271474, Vancouver, British Columbia
  - Royal Jubilee Hospital /ID# 271476, Victoria, British Columbia
  - Maritime Neurology /ID# 271867, Halifax, Nova Scotia
  - Neurocentre of Eastern Ontario /ID# 271865, Kingston, Ontario
  - Centricity /ID# 271477, London, Ontario
  - London Health Sciences Centre - Victoria Hospital & Children's Hospital /ID# 272031, London, Ontario
  - 360 Concussion Care /ID# 271972, Ottawa, Ontario
  - Bayshore Neurology /ID# 280213, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre /ID# 276844, Toronto, Ontario
  - Centre de Recherche St-Louis /ID# 272843, Lévis, Quebec
  - Genge Partners /ID# 273302, Montreal, Quebec
  - Diex Recherche Sherbrooke /ID# 271677, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-245